CLINICAL TRIAL: NCT05575739
Title: Evaluation of the Relationship Between the Psychological Level of Stress, Serum Oxidative Stress, Follicular Fluid Oxidative Stress, Ovarian Hormones and Response to Gonadotropin Stimulation During IVF (in Vitro Fertilisation) Procedures.
Brief Title: Evaluation of the Relationship Between Oxidative Stress and Human Reproduction
Acronym: OxidStressHR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Calla IVF Center (Other)
Responsible Party: Principal Investigator, Huniadi Anca Carmen, Dr., Calla IVF Center
Other Study IDs: CallaIVF
Record Dates: First submitted 2022-09-16; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: IVF; Pregnancy; Oxidative Stress; Fertility Disorders
Keywords: Oxidative Stress; In vitro fertilisation; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male factor: Couples that have just the male factor as cause of infertility
  Interventions: Diagnostic Test: Measurement of oxidative stress levels (Malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonylated proteins )
- Other causes of infertility: diminished ovarian reserve polycystic ovarian syndrome unexplained infertility tubal factor
  Interventions: Diagnostic Test: Measurement of oxidative stress levels (Malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonylated proteins )

INTERVENTIONS:
Diagnostic Test: Measurement of oxidative stress levels (Malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonylated proteins ) — Follicular fluid and serum were obtained within 1 hour of oocyte recovery. Considerable care was taken to pool follicular fluid uncontaminated with blood. The samples were processed by centrifuge and 1-mL aliquots stored ar -80ºC until assay. Malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonylated proteins were measured from follicular fluid and plasma according to manufacturer's protocol. This assay has been described as highly sensitive. Data were expressed as millimoles per liter from the reference curve.

SUMMARY:
The aim of the study is to investigate the role of oxidative stress in female infertility and the relationship between the stress as it is illustrated by questionnaires, serum markers, follicular fluid markers, and ovarian response in assisted reproduction.

DETAILED DESCRIPTION:
The investigators included patients that underwent an in vitro fertilization procedure in CALLA IVF Clinic.

All the patients had at least one ovarian stimulation cycle. In day two of the menstrual cycle the patients had a blood test for serum FSH(follicular stimulant hormone) E2 (estradiol) LH(Luteinizing hormone) and P(progesterone) as well as an ultrasound to asses the antral follicular count(AFC). The same day(day 2) the stimulation protocol begins. These four parameters are tested few times during the stimulation. The average stimulation protocol is 11 days. When the serum levels of hormones and ultrasound measurements of follicles reach the needed values (E2>1000pg/mL and follicles over 17mm) the hCG trigger is received. Transvaginal ultrasound guided oocyte retrieval was performed at 34-36 hours later. ICSI (intracitoplasmatic sperm injection) was performed and the fertilization by the presence of two pronuclei was confirmed 16-20 hours after the injection.

Follicular fluid and serum were obtained within 1 hour of oocyte recovery. Considerable care was taken to pool follicular fluid uncontaminated with blood. The samples were processed by centrifuge and 1-mL aliquots stored ar -80ºC until assay. Malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonylated proteins were measured from follicular fluid and plasma according to manufacturer's protocol. This assay has been described as highly sensitive. Data were expressed as millimoles per liter from the reference curve.

The parameters that are being observed are: number of oocytes, fertilisation rate and number of embryos.

ELIGIBILITY:
Inclusion Criteria:

* all patients with the Infertility diagnosis (trying to conceive for over 12 months having regular unprotected sexual intercourse) and having an ovarian puncture during an IVF procedure

Exclusion Criteria:

* patients that need sperm and egg donors
* patients that refuse being enrolled in the study

Ages: 20 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Population is homogeneous. Study group are females that struggle with infertility.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-14 (Estimated)

PRIMARY OUTCOMES:
Follicular fluid and serum: malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonated proteins on the day of ovarian puncture in in vitro fertilisation procedures. | 7 days (from ovulation trigger to day 5 embryo, meaning blastocyst)
  The primary outcome of the study is to establish the correlation between the oxidative stress markers and the ovarian response and the IVF(in vitro fertilization) success (number of oocytes retrieved, mature oocytes, fertilization rate, blastulation rate).
Correlation between the levels of oxidative stress markers (malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonated proteins) and the cause of infertility. | 7 days (from ovulation trigger to day 5 embryo, meaning blastocyst)
  The values of malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonated proteins in patients going trough an IVF procedure and the way the are associated with the cause of infertility. If the values differ between the two groups and if they impact the outcome of the IVF procedure (number of oocytes retrieved, mature oocytes, fertilization rate, blastulation rate) in either group.

SECONDARY OUTCOMES:
Questionnaire of psychological evaluation of perception of the day to day level of stress and the association with the levels of oxidative stress in the day of ovarian puncture. | 1-2 hours
  Perceived stress questionnaire - having 3 levels of stress according to the points in each question.
Correlation between maternal age and ovarian reserve and the values of oxidative stress markers (malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonated proteins) in the ovarian stimulation outcome. | 18 months
  The values of antimullerian hormone in ng/mL and the values of oxidative stress markers (malondialdehide, glutathione disulphate, total antioxidant capacity, superoxide dismutase and carbonated proteins) and the succes rate of the IVF procedure.
Correlation between HOMA-IR value (fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5), insulino-resistance and the body mass index, values of oxidative stress markers and ovarian stimulation outcome. | Day 1 of ovarian stimulation
  HOMA-IR value and body mass index in patients during the cycle of ovarian stimulation for IVF procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anca Huniadi, Study Chair — CALLA IVF
Locations (1):
- Calla Ivf, Oradea, Bihor County, Romania